CLINICAL TRIAL: NCT06741839
Title: Efficacy and Safety of Confocal Laser Endomicroscopy Guided Medical Thoracoscopy for the Diagnosis of Pleural Disease: a Multicenter Randomized Controlled Trial
Brief Title: Confocal Laser Endomicroscopy Guided Medical Thoracoscopy for the Diagnosis of Pleural Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Chief physician, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2022YFC2404404-3-1
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Pleural Diseases; Pleural Effusion
MeSH Terms: conditions — Pleural Diseases; Pleural Effusion

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nCLE guided biopsy (Experimental)
  Interventions: Procedure: Confocal laser endomicroscopy guided pleural biopsy using medical thoracoscopy
- Visual biopsy (Experimental)
  Interventions: Procedure: Plerual biopsy using medical thoracoscopy

INTERVENTIONS:
Procedure: Confocal laser endomicroscopy guided pleural biopsy using medical thoracoscopy — After the completion of the routine thoracoscopic examination, the biopsy location was determined based on the results of chest CT/ ultrasound. The benign and malignant states of pleural lesions were explored by nCLE and image records were collected. Then, the biopsy tissues were collected under the guidance of nCLE.
  Arms: nCLE guided biopsy
Procedure: Plerual biopsy using medical thoracoscopy — After the completion of the routine thoracoscopic examination, the biopsy location was determined according to the results of chest CT/ ultrasound, and random pathological biopsy was performed, and biopsy tissues were collected by biopsy forceps.
  Arms: Visual biopsy

SUMMARY:
A prospective multicenter randomized controlled trial was conducted to evaluate the efficacy and safety of thoracoscopic biopsy guided by confocal optical real-time microscopic imaging (nCLE) in the diagnosis of fibrinal pleurisy of unknown etiology. Patients with fibrinous pleurisy of unknown etiology who were to undergo thoracoscopic pleural biopsy were enrolled and informed consent was signed. Subjects were randomized to either the nCLE guided biopsy Group (Group A) or the visual biopsy group (Group B) according to the randomization table (1:1 ratio). nCLE was used to probe the benign and malignant status of pleural lesions, compare the consistency of random pathological biopsy or nCLE guided biopsy with histopathological results, compare whether nCLE guided biopsy can reduce the number of thoracoscopic biopsies, and follow up short-term postoperative complications to evaluate its safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral pleural effusion of unclear aetiology after less invasive means of diagnosis;
* Patients who intend to undergo a thoracoscopic pleural biopsy to determine the cause of pleural effusion;
* Sign informed consent.

Exclusion Criteria:

* There is an uncorrectable coagulation disorder or anticoagulation therapy that cannot be stopped before surgery;
* Hemodynamic instability;
* Refractory hypoxemia;
* Patients with pregnant and lactating patients
* Any illness or condition that interferes with the completion of the initial or subsequent assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of biopsies obtained for pathological diagnosis | 12 months

SECONDARY OUTCOMES:
Incidence of operation-related complications | 7 days
Diagnostic accuracy of pleural diseases | 12 months
time of operation | the day of operation
Overall diagnosis rate of pleural disease | 12 months

IPD SHARING:
Plan to Share IPD: No